CLINICAL TRIAL: NCT03086018
Title: A Comparative, Controlled, Clinical Investigation and Quality Control of a New Hearing Aid in Comparison to the Currently Marketed Device
Brief Title: A Comparative, Controlled, Clinical Investigation and Quality Control of a New Hearing Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernafon AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BF001-1611
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: A single group, controlled test design will be used. There are various aspects of testing including lab and field tests.
Masking Description: The hardware will be obviously different from the control devices and impossible to blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Successor hearing aid to Juna (Experimental): The intervention is the new device which is the successor to the Juna device. The participants will use their current device as a control. The will wear the intervention device for approximately two weeks.
  Interventions: Device: Successor hearing aid to Juna

INTERVENTIONS:
Device: Successor hearing aid to Juna — The participants will all be experienced hearing instrument device users and will be switched from their current (control) devices to the new test device which succeeds the Juna device.

SUMMARY:
The aim of this study is to investigate the performance of the hearing aid under laboratory as well as everyday conditions. In addition, the performance data of the hearing aid are compared with a Bernafon hearing aid already available on the market.

The hearing aids are adapted according to the user requirements. The data collected in the study is intended to show that the benefit of the hearing aid being examined is identical or better than the current CE-marked hearing aid. A further aim is to improve the adaptation of the hearing device in such a way that the benefit for people with hearing impairments can be increased.

DETAILED DESCRIPTION:
The reason for this study is to evaluate a new hearing aid. The goal is to evaluate the audiological performance and usability as well as features and functions in comparison to the hearing aid already CE marked. Furthermore, it is important to identify unexpected or unwanted behavior from the devices. This clinical investigation is a validation testing and is designed to evaluate the new hearing instrument system. As human subjects are involved, this validation test falls under the definition of a clinical investigation. The validation addresses the performance of the device with new functionality, and additionally addresses whether the end user can understand speech as well as with the current marketed device.

End users will be tested in the lab with speech tests and usability tests. They will also participate in field tests after which they will answer questionnaires concerning their experience with the instruments. Evaluating the overall performance of the hearing instrument is important to verify that the end user is satisfied with the device and that all user requirements are fulfilled. Many of the features available in the new device have already been validated and are used in devices currently on the market.

The purpose of this research is to show that the performance of the new device is as good as or better than the current device. Furthermore, speech should not be negatively affected with the addition of new features, the usability of the devices (that end users are able to handle the devices) should be as good as the current device, and there should be no artifacts or unwanted noises. Some measurements serve as quality control prior to product launch.

ELIGIBILITY:
Inclusion Criteria:

* All classifications of hearing loss (sensorineural, conductive, mixed)
* If the hearing loss is conductive or mixed it must be approved for amplification by a physician
* All shapes of hearing loss (flat, sloping, reverse slope, notch)
* Severity ranging from mild to severe
* German speaking
* Ability and willingness to sign the consent form

Exclusion Criteria:

* Contraindications for amplification
* Active ear disease
* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia, or other cognitive problems of the participant,
* A reduced mobility making them unable to attend weekly study appointments
* A reduced ability to describe auditory impressions and the usage of the hearing aids
* Uncooperative so that it is not possible to record a valid pure tone audiogram
* A strongly reduced dexterity
* Central hearing disorders
* Bernafon employees
* Family members of Bernafon employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Simon, AuD, Principal Investigator — Bernafon AG
Locations (1):
- Bernafon AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Successor Hearing Aid to Juna: The intervention is the new device which is the successor to the Juna device. The participants will use their current device as a control. They will wear the intervention device for approximately two weeks.
Period: Field Testing
Arm/Group | Experimental: Successor Hearing Aid to Juna
Started | 30
Completed | 30
Not Completed | 0
Period: Final Testing for End of Trial
Arm/Group | Experimental: Successor Hearing Aid to Juna
Started | 30
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: For this study all data gathered had to be included in the analysis. This means that some data is analyzed from 30 participants and some from only 28 for any data not gathered after the two participants dropped from the study.
Groups:
- Experimental: Successor Hearing Aid to Juna: The intervention is the new hearing aid which is the successor to the Juna device. The participants will use their current device as a control. They will wear the intervention device for approximately two weeks.
Arm/Group | Experimental: Successor Hearing Aid to Juna
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 67 [38 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 30
Hearing Instrument Experience [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility Performance
Description: Speech test scores will be measured with speech reception thresholds (SRTs) of speech in noise in three conditions: unaided, aided with the current device, and aided with the new device. The score is measured by the the signal-to-noise ratio (SNR) at which 50% of words in a sentence list are correctly repeated. The speech is always presented at 65 dB and the background noise varies to maintain the 50% correct. A lower SNR score indicates a better score. The maximum score will be 15 dB and the minimum will be -5 dB.
Time Frame: 2 hour period of speech testing during a lab appointment after wearing the devices for approximately 2 weeks.
Measure: Mean (Standard Deviation); unit: dB SNR
Arm/Group | Successor Hearing Aid to Juna
Number analyzed (Participants) | 28
dB SNR
  Unaided | -1.25 (1.45)
  Aided with current device | -3.89 (0.99)
  Adided with new device | -5.22 (1.09)

2. Secondary Outcome: Subjective Performance of Aided Benefit
Description: The subjective performance for the new device will be measured with the APHAB questionnaire (Abbreviated Hearing Aid Benefit Profile). The questionnaire is a list of 24 statement that the subjects must agree or disagree with using a scale of units from A to G (A being Always and G being Never). Each letter has a corresponding score used for the calculation: A receives 99, B receives 87, C receives 75, D receives 50, E receives 25, F recevies 12, and G receives 1.
  An average for each subscale is calculated, and a global or overall score can be calculated by taking the mean of the three positive subscales (Ease of communication, Background noise, and Reverberation). For these three subscales a higher score indicates a better performance. The highest possible score is 99 and the lowest is 1. The fourth scale (Aversiveness) is a negative scale meaning that a higher score means a worse performance. The highest possible score is 99 and the lowest is 1.
Time Frame: A 2 week time period during which they will wear the devices and answer questionnaires about the experience.
Population: For this questionnaire, two participants had left the study and data was not collected.
Measure: Median (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental: Successor Hearing Aid to Juna
Number analyzed (Participants) | 28
Units on a scale
  Ease of Communication | 37.38 (24.11)
  Background Noise | 44.29 (16.89)
  Reverberation | 42.08 (23.96)
  Aversiveness | -17.63 (26.14)
  Global Score | 40.30 (20.49)

3. Secondary Outcome: Speech Intelligibility Performance With New Feature
Description: Word recognition test scores will be measured with two signal-to-noise ratio (SNR) levels in percent correct in two conditions, with the new feature on and the new feature off.
  The test is a speech test with the words stated in noise at either a 5 dB SNR or a 15 dB SNR. The subject is presented with 5 rhyming words and must choose which word they heard. It is a forced choice meaning that the test will not continue with the next word until they've made a selection. They cannot leave any blank and are not penalized for wrong answers. The score is a percentage of words correct with the maximum score being 100% and the minimum being 0%. A higher score means a better outcome.
Time Frame: 2 hour period of speech testing during a lab appointment after wearing the devices for approximately 2 weeks.
Measure: Mean (Standard Deviation); unit: percent correct out of 100%
Arm/Group | Experimental: Successor Hearing Aid to Juna
Number analyzed (Participants) | 30
percent correct out of 100%
  +5 SNR WAKO Feature on | 73.5 (5.2)
  +5 SNR WAKO Feature off | 73.7 (4.95)
  +15 SNR WAKO Feature on | 87.27 (4.08)
  +15 SNR WAKO Feature off | 88.1 (4.63)

4. Secondary Outcome: Handling/Usability Performance
Description: The usability of the new device will be measured with a 3-point rating scale used by the tester to evaluate tasks performed by the end user as well as questionnaires and interviews.
  The questionnaire asks subjects to perform tasks, and the clinician rates the ease with which they complete the tasks. 2 is the highest score meaning that they could complete without help, 1 means that they required some assistance, and 0 means that they could not complete the task. A higher score means a better outcome.
Time Frame: 2 hour period of usability testing with tasks and questionnaires.
Measure: Number; unit: percentage of tasks scored with 2
Arm/Group | Experimental: Successor Hearing Aid to Juna
Number analyzed (Participants) | 30
percentage of tasks scored with 2 | 97

5. Secondary Outcome: Events
Description: Events will be measured by the reporting of unexpected sounds or behavior of the device through questionnaires, diaries, and interviews. The number of events reported including AEs related to the device will be used to measure the outcome. Less events is a better outcome.
Time Frame: A 2 hour period of interviews and questionnaires after having worn the devices for approximately 2 weeks and keeping a diary to make notes of device behavior.
Measure: Number; unit: Units of AEs related to device
Groups:
- Experimental: Succssor Hearing Aid to Juna: The intervention is the new device which is the successor to the Juna device. The participants will use their current device as a control. They will wear the intervention device for approximately two weeks.
Arm/Group | Experimental: Succssor Hearing Aid to Juna
Number analyzed (Participants) | 30
Units of AEs related to device | 4

ADVERSE EVENTS:
Time Frame: 4 months
Description: All Cause Mortality is not a separate item in the definition of adverse events used in the study. This is considered part of the serious adverse events definition. We identified two categories, Serious adverse events and Adverse Events. All events fall into one of these categories, so when it is not considered a serious adverse event, it is an adverse event.
Arm/Group | Experimental: Successor Hearing Aid to Juna
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Successor Hearing Aid to Juna (N=30)
Hospitalization due to accident (Social circumstances) | 1 (1) — Was hospitalized after an accident at home, in which the back was injured requiring surgery. Participant could not continue in trial. No causality to IMD
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Successor Hearing Aid to Juna (N=30)
Cold (General disorders) | 2 (3) — Two participants reported colds during the study. One of the two participants reported it twice (on two separate Occasions). No causality to IMD
Tore Meniscus (General disorders) | 1 (1) — Participant tore left meniscus when the foot was twisted while walking. No causality to IMD
Scratch on ear canal (General disorders) | 1 (1) — Participant reported discomfort in ear. Upon inspection, a small scratch was found on the ear canal.
Dome in Ear (Product Issues) | 1 (1) — Dome fell off in the ear canal.
Headache (General disorders) | 1 (1) — Participant reported getting a headache after being in too much noise
Irritation in ear (General disorders) | 1 (1) — Participant reported irritation and pain in ear after wearing the domes for a few days. Removed device till problem resolved.
Sore Concha (Product Issues) | 1 (1) — Sore spot in concha, which resolved overnight after removing the device for the evening.
Back Pain (General disorders) | 1 (1) — Trouble with lower back pain. No causality to IMD
Pressure point (General disorders) | 1 (2) — Pressure point in ear when device not in ear correctly. Problem resolved after removal of device.
Tore Groin muscle (General disorders) | 1 (1) — Tore groin muscle on the right side after picking up grandchild. No causality to IMD
Leg problem (General disorders) | 1 (1) — Leg problems caused by spinal cord compression. No causality to IMD
Face Swelling (General disorders) | 1 (1) — Face swelling caused by allergic reaction to eye drops. No causality to IMD

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT03086018/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT03086018/SAP_001.pdf